CLINICAL TRIAL: NCT07370662
Title: Effect of Resistance Exercises and Relaxation Therapy on Physical Function and Quality Of Life in Patients With Chronic Kidney Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rashid Latif Medical College (Other)
Responsible Party: Principal Investigator, Tahir Mahmood, Assistant Professor, Rashid Latif Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB/2024/159
Record Dates: First submitted 2026-01-19; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Kidney Disease (Mild to Moderate)
Keywords: Chronic Kidney Disease; Physical Function; Quality of Life; Resistance Exercises.; Relaxation Therapy
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Group A: Resistance exercises and relaxation therapy Group B: Resistance exercises, where Resistance exercise (knee and hip flexion and extension, and elbow extension)
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor was kept blind. The individuals measuring or evaluating a study's results, assessor was not aware of treatment group (intervention) a participant belongs to, preventing their expectations or biases from influencing the outcome measurement and ensuring more objective results.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resistance exercises (Active Comparator): Resistance exercise (knee and hip flexion and extension ,and elbow extension)
  Interventions: Other: Resistance exercises:
- Relaxation exercise (Experimental): Diaphragmatic Breathing + Pursed Lip Breathing
  Interventions: Other: Resistance exercises:; Other: Relaxation exercise

INTERVENTIONS:
Other: Resistance exercises: — The researcher taught patients this exercise and encouraged them to do it daily each once about 20 to 30 minutes. The exercise started with moderate intensity of no more than 10 minutes then time of practice increased gradually to 30 minutes. Resistance exercise included the following: Knee and hip flexion and extension, elbow extension. The repetition was be 15-20 times
Other: Relaxation exercise — Relaxation exercise (diaphragmatic breathing, pursed lip breathing) Diaphragmatic breathing is intended to help patient use the diaphragm correctly while breathing to strengthen the diaphragm and decrease the work of breathing. Patient was instructed to sit comfortably with the knees bent and the shoulders, head and neck relaxed. Breathe in slowly through the nose so that the stomach moves out against the hand. Then exhaled through pursed lib technique so that stomach moves in again. Patients was instructed to place one hand on the upper chest and the other just below the rib cage. This was allowing patient to feel the diaphragm move as he or she breathe. Patients was instructed to practice this exercise 5-10 minutes about 3-4 times per day.
  Arms: Relaxation exercise

SUMMARY:
The significance of this study to compare the effect of resistance exercises and relaxation therapy to find out which technique is more effective for improving physical function and quality of life in chronic kidney disease patient.

The study was aimed to determine the effect of resistance exercises and relaxation therapy on physical function and quality of life in patients with chronic kidney disease.

We hypothesized if there was significant effect of resistance exercises and relaxation therapy on physical function and quality of life in patients with chronic kidney disease.

Group A: Relaxation therapy and Resistance exercises. Group B: Resistance exercises.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a pathophysiological process, where the kidneys experience a slow, progressive and irreversible decline in function where the body's ability fail in maintaining metabolism and fluid and electrolyte balance causes the occurrence of uremia.

Individuals of all ages and both sexes benefit from moderate-intensity physical activity, with diminished risk of cardiovascular diseases, maintenance of muscle strength, fewer symptoms of depression and anxiety and improved quality of life. Resistance exercises, alone and in combination with other exercises have shown beneficial outcomes in improving physical fitness, walking capacity, cardiovascular outcomes, and health-related quality of life (HRQoL). However, relaxation techniques are considered successful in improving the condition of patients. Deep breathing relaxation techniques can reduce oxidative stress, increase cellular energy, increase elasticity of blood vessels and improve circulation, so that the final result can reduce and even overcome fatigue. The technique is easy to do, easy to learn, does not harm and a less costs is the advantage of deep breathing relaxation techniques. Resistance training has been successfully recommended as a method of gaining lean mass, strength and physical functioning in frail elderly persons and those with chronic diseases, including patients with cardiovascular and kidney diseases

ELIGIBILITY:
Inclusion Criteria:

* Age (30-65years).
* Both Male and female.
* Patient able to stand and walk independently.
* Patient with mild to moderate stage of chronic kidney disease.

Exclusion Criteria:

* Physical disability.
* Acute Myocardial infarction.
* Kidney transplant.
* Pregnant women.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2024-08-12 (Actual); Primary Completion 2025-03-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
SF 36 (Quality of Life) | Pre-test (Baseline) and Post-test (08 Weeks)
  To assess patients Quality of life SF-36 was used. It provides information on 8 scales, scoring from0(worst health) to100(best health), and on the physical component scale (PCS) and the mental component scale (MCS), normalized scores representing overall physical and mental functioning

SECONDARY OUTCOMES:
Sit-to-Stand test | Pre-test (Baseline) and Post-test (08 Weeks)
  The STS 10 consisted of measuring the seconds employed by the patient to stand up from the sitting position, and to sit down for 10 consecutive times as quickly as possible. STS-10 is proved to be a feasible measure to detect changes resulting from an exercise intervention [ After 5 minutes for recuperation, the patient performed the STS 60 consisting of standing-up from a chair and sitting-down again as many times as possible during a 60 second time period.
6-minute walk test | Pre-test (Baseline) and Post-test (08 Weeks)
  It was used as an indicator of patients' exercise capacity. The total distance covered by subjects during 6 minutes on a walk of 20 meters in length along an internal corridor of the HD unit was recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Arif memorial teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
The data will be shared on reasonable request

REFERENCES:
- [Background] Segura-Ortí E, Kouidi E, Lisón J. Effect of resistance exercise during hemodialysis on physical function and quality of life: randomized controlled trial. Clinical nephrology. 2009;71(5):527.
- [Background] Barcellos FC, Santos IS, Mielke GI, Del Vecchio FB, Hallal PC. Effects of exercise on kidney function among non-diabetic patients with hypertension and renal disease: randomized controlled trial. BMC nephrology. 2012;13:1-7.
- [Background] Abd Elbaky M, Zaki S, Amin N, Ali R. Impact of Intradialytic Rehabilitation Program on General Health of Chronic Kidney Disease Patients. American Journal of Nursing. 2018;6(5):263-72